CLINICAL TRIAL: NCT06204211
Title: Genetic Research on High Myopic Individuals in Northern China
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Liping Du, Professor, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2022-KY-0512-002
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: High Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood DNA were isolated utilizing the QIAamp DNA Blood Mini Kit (Qiagen, Hilden, North Rhine-Westphalia, Germany). And subsequently, the purity and concentration of obtained DNA were surveyed by the Nanodrop 2000 spectrophotometer (Thermo Fisher Scientific, Wilmington, Delaware, the United States of America), after which the normalization of qualified DNA samples followed. Finally, standardized DNA specimens were hold at -80 ℃ for future use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High myopia: HM participants characterized by AL ≥ 26.00 mm or SE ≤ -6.00 D in at least one eye at the Department of Ophthalmology of the First Affiliated Hospital of Zhengzhou University (Zhengzhou, Henan Province, China) from May 2022 to April 2023 are included as cases.
  Interventions: Diagnostic Test: ophthalmologic examinations
- Control: Demographic-matched emmetropic volunteers without consanguinity serve as controls.
  Interventions: Diagnostic Test: ophthalmologic examinations

INTERVENTIONS:
Diagnostic Test: ophthalmologic examinations — All the included personnel underwent routine ophthalmologic examinations on binoculus, including slit lamp microscope observation, intraocular pressure, diopters of refractive error, best corrected visual acuity, AL measurement, fundus photography and optical coherence tomography, adhering to the established and normalized principles.

SUMMARY:
HM, which can dramatically cripple the eyesight of those affected, is a rampant ophthalmic disorder around the globe. It is in recent years that substantial studies covering the relationship between distinct variations and HM susceptibility sprang expeditiously. However, these studies have not yielded sufficiently credible and universally significant conclusions. Consequently, the study is conducted by including HM subjects residing in Northern China to explicitly illustrate this issue.

DETAILED DESCRIPTION:
As a serious pattern of myopia, high myopia (HM) generally refers to a condition where the spherical equivalent (SE) refraction exceeds -6.00 diopters (D) or the axial length (AL) is longer than 26.00 mm. Abundant studies have indicated the strong correlation of HM with multiple vision-threatening ophthalmic diseases, including rhegmatogenous retinal detachment, retinoschisis, retinochoroid atrophy and open-angle glaucoma. It is reported that the worldwide prevalence of HM has surpassed over 2.9% in recent years. And a study on subjects living in Minnesota from the 1960s to the 2010s demonstrates that the data has progressively increasing from 2.8% to 8.3%, which is not related with gender or race, although no evident significance has yet been proved in some groups. What's worse, it is speculated that HM patients are expected to account for 9.8% of the global population by 2050, which will gravely hinder the progress of social development. As a result, it is of profound implications to explore the pathogenesis of HM and the prospective therapeutic or remedial strategies.

What has been universally acknowledged is that both environmental and genetic factors matter much in the onset and exacerbation of myopia, with the latter particularly predominating in the etiology of HM. Accordingly, discussing the causation of HM from heredity version is likely to be the most promising research field, which is just the researchers' interest at the present.

ELIGIBILITY:
Inclusion Criteria:

* HM participants are characterized by AL ≥ 26.00 mm or SE ≤ -6.00 D in at least one eye.

Exclusion Criteria:

* Individuals with other ocular or systemic connective tissue diseases were excluded.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The gender of subjects is divided according to the reports of Heidari et al (see the reference 1).
Study Population: We enrolled HM participants characterized by AL ≥ 26.00 mm or SE ≤ -6.00 D in at least one eye at the Department of Ophthalmology of the First Affiliated Hospital of Zhengzhou University (Zhengzhou, Henan Province, China) from May 2022 to April 2023 as cases and unrelated normal volunteers with SE ranging from -0.50 D to +0.50 D as controls.
Sampling Method: Probability Sample
Enrollment: 1340 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
diopter | 1 hour
  This study performs the subgroup analysis based on SE (≤ -20.00 D, -20.00 ~ -15.00 D, -15.00 ~ -10.00 D, and -10.00 ~ -6.00 D) to clarify the correlation between different genetic SNPs and HM inclination more thoroughly.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Du, Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Liping Du, Zhengzhou, Henan, China

REFERENCES:
- [Background] Heidari S, Babor TF, De Castro P, Tort S, Curno M. Sex and Gender Equity in Research: rationale for the SAGER guidelines and recommended use. Res Integr Peer Rev. 2016 May 3;1:2. doi: 10.1186/s41073-016-0007-6. eCollection 2016. PMID 29451543
- [Derived] Gao W, Zhang M, An G, Yang F, Li L, Jin X, Du L. The association of ARR3 genetic polymorphisms with pathologic myopia in Northern Chinese population. Exp Eye Res. 2025 Dec;261:110691. doi: 10.1016/j.exer.2025.110691. Epub 2025 Oct 9. PMID 41076047